CLINICAL TRIAL: NCT02377752
Title: A Phase 1 Study of Olaratumab in Japanese Patients With Advanced Soft Tissue Sarcoma or Advanced Solid Tumors
Brief Title: A Study of Olaratumab in Japanese Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15678; I5B-JE-JGDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — olaratumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A cohort 1: Olaratumab+Doxorubicin (Experimental): 15 milligram per kilogram (mg/kg) of olaratumab administered intravenously (IV) on Day 1 and Day 8, and 25 milligram per square meter (mg/m2) of doxorubicin administered IV on Day 1, Day 2, and Day 3 every 21-day cycle for up to 6 cycles or until the cumulative dose of doxorubicin reached 500 mg/m2, whichever came later, followed by 15 mg/kg of olaratumab IV monotherapy on Day 1 and Day 8 in subsequent cycles. Participants may continue to receive treatment until discontinuation criteria are met
  .
  Interventions: Biological: Olaratumab; Drug: Doxorubicin
- Part A cohort 2: Olaratumab+Doxorubicin (Experimental): 15 mg/kg of olaratumab administered IV on Day 1 and Day 8, and 75 mg/m2 of doxorubicin administered IV on Day 1 every 21 day-cycle for up to 6 cycles or until the cumulative dose of doxorubicin reached 500 mg/m2, whichever came later, followed by 15 mg/kg of olaratumab IV monotherapy on Day 1 and Day 8 in subsequent cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Biological: Olaratumab; Drug: Doxorubicin
- Part A cohort 3 Olaratumab + Doxorubicin (Experimental): 20 mg/kg loading dose of olaratumab administered IV on Day 1 and Day 8 in Cycle 1, followed by 15 mg/kg IV on Day 1 and Day 8 in subsequent cycles, and 75 mg/m2 of doxorubicin administered IV on Day 1 of every 21 day-cycle up to 6 cycles or until the cumulative dose of doxorubicin reached 500 mg/m2, whichever came later, followed by 15 mg/kg of olaratumab IV monotherapy on Day 1 and Day 8 in subsequent cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Biological: Olaratumab; Drug: Doxorubicin
- Part B: Olaratumab (Experimental): 15 mg/kg olaratumab administered IV on Day 1 and Day 8 of every 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Biological: Olaratumab

INTERVENTIONS:
Biological: Olaratumab — Administered IV
  Other Names: LY3012207; IMC-3G3
Drug: Doxorubicin — Administered IV
  Arms: Part A cohort 1: Olaratumab+Doxorubicin; Part A cohort 2: Olaratumab+Doxorubicin; Part A cohort 3 Olaratumab + Doxorubicin

SUMMARY:
This study consists of 2 parts (Part A and Part B). The main purpose of Part A is to evaluate safety and side effects of olaratumab in combination with doxorubicin in Japanese participants with a group of rare cancers (advanced solid tumors, especially advanced soft tissue sarcoma [STS].) The main purpose of Part B is to evaluate how much olaratumab gets into the blood stream of Japanese participants with advanced solid tumors and how long it takes the body to get rid of it.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Have histological or cytological evidence of a diagnosis of advanced or metastatic solid tumor, especially STS, which is not amenable to treatment with surgery or radiotherapy. Part B: Have histological or cytological evidence of a diagnosis of solid tumor that is advanced or metastatic.
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).
* Have given written informed consent prior to any study-specific procedures.
* Have adequate organ and coagulation function
* Have an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of less than or equal to 1.
* Have discontinued previous treatments for cancer and recovered from the acute effects of therapy.
* (Part A only) Have a prestudy echocardiogram with an actual left ventricular ejection fraction greater than or equal to 50%, within 21 days prior to first dose of study medication.
* All participants agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following last dose of study drug.
* Female participants:

  * must either be women not of child-bearing potential due to surgical sterilization confirmed by medical history, or menopause or
  * women of child-bearing potential who test negative for pregnancy within 7 days before the first dose of study drug based on serum or urine pregnancy test and agree not to breast feed during the study and for 3 months following the last dose of the study drug(s)
* Have an estimated life expectancy of more than or equal to 3 months in the judgment of the investigator.

Exclusion Criteria:

* Have received treatment within 21 days of the initial dose of study drug with an investigational product or non-approved use of a drug or device for non-cancer indications or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* (Part A only) Have received prior treatment with doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones
* (Part A only) Have received prior radiation therapy to the mediastinal/pericardial area.
* Have symptomatic central nervous system malignancy or metastasis. Participants with treated central nervous system (CNS) metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 60 days.
* Have an elective or a planned major surgery to be performed during the course of the study.
* Have an uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure greater than class II of the New York Heart Association guideline, severe myocardial insufficiency, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 6 months prior to study entry.
* Have a known allergy to any of the treatment components.
* Have a history of allergic reactions attributed to compounds of chemical or biologic composition similar to that of olaratumab.
* Have a known active fungal, bacterial, and/or known viral infection
* Have a corrected QT interval of greater than 470 milliseconds (msec) on screening electrocardiogram (ECG)
* Have a second primary malignancy that, in the judgment of the investigator and sponsor, may affect the interpretation of results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Kōtoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Suita-shi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered to have competed the study if the study discontinued due to adverse event, progressive disease (PD) or withdrawal by subject.
Groups:
- Part A Cohort 1: Olaratumab+Doxorubicin: 15 milligram per kilogram (mg/kg) of olaratumab administered intravenously (IV) on Day 1 and Day 8, and 25 milligram per square meter (mg/m2) of doxorubicin administered IV on Day 1, Day 2, and Day 3 every 21-day cycle for up to 6 cycles or until the cumulative dose of doxorubicin reached 500 mg/m2, whichever came later, followed by 15 mg/kg of olaratumab IV monotherapy on Day 1 and Day 8 in subsequent cycles. Participants may continue to receive treatment until discontinuation criteria are met
Period: Overall Study
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin | Part B: Olaratumab
Started | 7 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 7 | 6 | 6 | 6
Completed | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received any amount of study drugs (either olaratumab or doxorubicin) in Part A and Part B.
Groups:
- Part A Cohort 1: Olaratumab+Doxorubicin: 15 mg/kg of olaratumab administered IV on Day 1 and Day 8, and 25 mg/m2 of doxorubicin administered IV on Day 1, Day 2, and Day 3 every 21-day cycle for up to 6 cycles or until the cumulative dose of doxorubicin reached 500 mg/m2, whichever came later, followed by 15 mg/kg of olaratumab IV monotherapy on Day 1 and Day 8 in subsequent cycles. Participants may continue to receive treatment until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin | Part B: Olaratumab | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (15.3) | 45.8 (11.0) | 40.7 (8.7) | 59.3 (8.1) | 49.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 5 | 16
  Male | 3 | 4 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 6 | 6 | 6 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 6 | 6 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Clinically significant events were defined as serious adverse events (SAE). A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to Study completion (Up To 3.5 Years)
Population: All enrolled participants who received any amount of study drugs (either olaratumab or doxorubicin) in Part A.
Measure: Number; unit: participants
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 7 | 6 | 6
participants | 1 | 4 | 1

2. Primary Outcome: Part A: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is defined as adverse event (AE) during Cycle 1 (Days 1 through 21) that was possibly related to the study drug and toxicities considered by the investigator as dose limiting. A summary of other nonserious AEs, and all serious adverse events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Cycle 1 (21 Days)
Population: All enrolled patients who completed Cycle 1 (initial 21-day treatment period), or who discontinued due to DLT during Cycle 1 in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 7 | 6 | 6
Participants | 0 | 1 | 0

3. Primary Outcome: Part B: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Olaratumab
Description: Maximum observed serum concentration (Cmax) of olaratumab is reported.
Time Frame: Cycle (C) 1 Day (D) 1 and C3 D1: Pre-infusion, Immediately postinfusion and 1, 24, 48, 72 and 168 hours (h) postinfusion; C1 D8 and C3 D8: Pre- infusion, Immediately postinfusion and 1, 48, 72, 168 and 336 h postinfusion
Population: All enrolled participants who received any amount of study drug (olaratumab) and had evaluable pharmacokinetics (PK) data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Part B: Olaratumab
Number analyzed (Participants) | 6
microgram per milliliter (μg/mL)
  Cycle 1 Day 1 | 322 (22)
  Cycle 1 Day 8 | 409 (32)
  Cycle 3 Day 1: number analyzed (Participants) | 3
  Cycle 3 Day 1 | 396 (16)
  Cycle 3 Day 8: number analyzed (Participants) | 3
  Cycle 3 Day 8 | 478 (15)

4. Primary Outcome: Part B: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of Olaratumab
Description: AUC(0-t) hours (h), area under the serum concentration versus time curve from time zero to t hours at AUC(0-168h) for Cycle 1 Day 1 and Cycle 3 Day 1, AUC(0-336h) for Cycle 1 Day 8 and Cycle 3 Day 8 of Olaratumab is reported.
Time Frame: as for outcome 3
Population: All enrolled participants who received any amount of study drug (olaratumab) and had evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/mL (μg*h/mL)
Arm/Group | Part B: Olaratumab
Number analyzed (Participants) | 6
microgram*hour/mL (μg*h/mL)
  Cycle 1 Day 1: AUC(0-168h) | 23300 (26)
  Cycle 1 Day 8: AUC(0-336h): number analyzed (Participants) | 5
  Cycle 1 Day 8: AUC(0-336h) | 48100 (47)
  Cycle 3 Day 1: AUC(0-168h): number analyzed (Participants) | 3
  Cycle 3 Day 1: AUC(0-168h) | 39800 (14)
  Cycle 3 Day 8: AUC(0-336h): number analyzed (Participants) | 2
  Cycle 3 Day 8: AUC(0-336h) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of AUC(0-336h) = 66500 μg*h/mL, 92300 μg*h/mL.

5. Secondary Outcome: Part A: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Olaratumab
Description: Maximum observed serum concentration (Cmax) of olaratumab is reported.
Time Frame: Cycle (C) 1 Day (D) 1 and C3 D1: Pre-infusion, Immediately postinfusion and 1.5, 24, 48, 72 and 168 hours (h) postinfusion; C1 D8 and C3 D8: Pre- infusion, Immediately postinfusion and 1, 48, 72, 168 and 336 h postinfusion
Population: All enrolled participants who received any amount of study drugs (either olaratumab or doxorubicin) and had evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 6 | 6 | 6
microgram per milliliter (μg/mL)
  Cycle 1 Day 1 | 274 (30) | 301 (25) | 470 (27)
  Cycle 1 Day 8 | 353 (40) | 351 (20) | 610 (33)
  Cycle 3 Day 1: number analyzed (Participants) | 4 | 4 | 5
  Cycle 3 Day 1 | 351 (28) | 390 (13) | 545 (34)
  Cycle 3 Day 8: number analyzed (Participants) | 4 | 4 | 5
  Cycle 3 Day 8 | 415 (28) | 474 (13) | 541 (41)

6. Secondary Outcome: Part A: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of Olaratumab
Description: as for outcome 4
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*h/mL)
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 6 | 6 | 6
microgram*hour per milliliter (μg*h/mL)
  Cycle 1 Day 1: AUC(0-168h) | 21700 (36) | 21900 (25) | 34300 (29)
  Cycle 1 Day 8: AUC(0-336h) | 47300 (32) | 42000 (36) | 74100 (42)
  Cycle 3 Day 1: AUC(0-168h): number analyzed (Participants) | 4 | 4 | 5
  Cycle 3 Day 1: AUC(0-168h) | 33600 (31) | 36000 (15) | 42500 (51)
  Cycle 3 Day 8: AUC(0-336h): number analyzed (Participants) | 4 | 4 | 5
  Cycle 3 Day 8: AUC(0-336h) | 63000 (28) | 68400 (15) | 77700 (68)

7. Secondary Outcome: Part A: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Doxorubicin
Description: Maximum observed plasma concentration (Cmax) of doxorubicin is reported.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 3, Cycle 3 Day 1, Cycle 3 Day 2 and Cycle 3 Day 3: Immediately postinfusion
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin
Number analyzed (Participants) | 6
nanogram/milliliter (ng/mL
  Cycle 1 Day 1 | 594 (86)
  Cycle 1 Day 2: number analyzed (Participants) | 5
  Cycle 1 Day 2 | 444 (97)
  Cycle 1 Day 3: number analyzed (Participants) | 4
  Cycle 1 Day 3 | 384 (105)
  Cycle 3 Day 1: number analyzed (Participants) | 3
  Cycle 3 Day 1 | 855 (29)
  Cycle 3 Day 2: number analyzed (Participants) | 4
  Cycle 3 Day 2 | 742 (45)
  Cycle 3 Day 3: number analyzed (Participants) | 4
  Cycle 3 Day 3 | 884 (24)

8. Secondary Outcome: Part A: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Doxorubicin
Description: Maximum observed plasma concentration (Cmax) of doxorubicin is reported.
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1: Immediately postinfusion, 0.5, 1, 2, 4, 8, 24, 48, and 72 h postinfusion
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 6 | 6
nanogram/milliliter (ng/mL)
  Cycle 1 Day 1 | 2660 (25) | 2790 (12)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 3 Day 1 | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 1791.71 ng/mL, 1812.61 ng/mL. | 2900 (19)

9. Secondary Outcome: Part A: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of Doxorubicin
Description: Area under the concentration verses time curve from zero to infinity (AUC[0-∞]) of doxorubicin is reported.
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1: Immediately postinfusion, 0.5, 1, 2, 4, 8, 24, 48, and 72 h postinfusion
Population: All enrolled participants who received any amount of study drugs (either olaratumab or doxorubicin) and had evaluable PK data in Part A. AUC data is not available for Part A cohort 1 as PK was evaluated immediately post infusion of doxorubicin in Part A cohort 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Arm/Group | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin
Number analyzed (Participants) | 6 | 6
nanogram*hour/mL (ng*h/mL)
  Cycle 1 Day 1 | 3070 (12) | 3020 (15)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 3 Day 1 | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of AUC[0-∞] = 2990 ng*h/mL, 3410 ng*h/mL. | 3720 (17)

10. Secondary Outcome: Change From Baseline in Percentage of Participants With a Tumor Response
Description: Tumor response was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1. Complete Response (CR) is disappearance of all target lesions; Partial Response (PR) is greater than or equal to (≥) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to Study completion (Up To 3.5 Years)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin | Part B: Olaratumab
Number analyzed (Participants) | 7 | 6 | 6 | 6
percentage of participants | 0 [0.0 to 35.4] | 33.3 [9.7 to 70.0] | 33.3 [9.7 to 70.0] | 0 [0.0 to 39.0]

ADVERSE EVENTS:
Time Frame: Baseline to Study completion (Up To 3.5 Years)
Description: All enrolled participants who received any amount of study drugs (either olaratumab or doxorubicin) in Part A and Part B.
Arm/Group | Part A Cohort 1: Olaratumab+Doxorubicin | Part A Cohort 2: Olaratumab+Doxorubicin | Part A Cohort 3 Olaratumab + Doxorubicin | Part B: Olaratumab
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/6 | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Olaratumab+Doxorubicin (N=7) | Part A Cohort 2: Olaratumab+Doxorubicin (N=6) | Part A Cohort 3 Olaratumab + Doxorubicin (N=6) | Part B: Olaratumab (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Olaratumab+Doxorubicin (N=7) | Part A Cohort 2: Olaratumab+Doxorubicin (N=6) | Part A Cohort 3 Olaratumab + Doxorubicin (N=6) | Part B: Olaratumab (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (5) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 3 (4) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (9) | 6 (11) | 6 (8) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 4 (5) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 5 (5) | 3 (3) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 4 (6) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 3 (4) | 4 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 3 (3) | 3 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (8) | 5 (14) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (9) | 6 (13) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (6) | 2 (3) | 4 (5) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 3 (5) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 6 (6) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators are fully restricted to publish any results of the study without sponsor's permission.

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02377752/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT02377752/SAP_001.pdf